CLINICAL TRIAL: NCT02684344
Title: Prophylactic Tamsulosin Use for Prevention of Post-Operative Urinary Retention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Edward Messing, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 59730
Record Dates: First submitted 2016-02-08; First posted 2016-02-18 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Post-Operative Urinary Retention
Keywords: Post-Operative Urinary Retention
MeSH Terms: interventions — Tamsulosin; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tamsulosin Group (Experimental): Subjects will receive:
  1. 0.4mg tamsulosin by mouth nightly for 3 doses prior to the day of surgery and for 2 doses following surgery
  2. education about signs and symptoms of urinary retention
  Interventions: Drug: Tamsulosin; Other: Education
- Education Group (Active Comparator): Subjects will receive:
  1) education about signs and symptoms of urinary retention
  Interventions: Other: Education

INTERVENTIONS:
Drug: Tamsulosin — Tamsulosin may have prophylactic properties against post-operative urinary retention
  Other Names: Flomax
  Arms: Tamsulosin Group
Other: Education — Education about signs and symptoms of urinary retention

SUMMARY:
This randomized open-label study will be comprised of 2 cohorts: one control group and one treatment group. The trial will be conducted as an open label randomized trial to evaluate the efficacy of tamsulosin in the prevention of post-operative urinary retention. The study will include pre- and post-surgical evaluations of patients including symptoms of urinary retention and any adverse effects contributable to the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Any male age 40 or older
* Scheduled to undergo one of the planned surgeries (thoracic, general, or urologic)
* Ability to give informed consent

Exclusion Criteria:

* Current use of alpha blocker
* Current use of a strong CYP 3A4 inhibitors
* Any allergy to tamsulosin, alpha-blocker medication class, or anaphylaxis allergy to sulfate containing medications
* Patients with any upcoming surgery for cataracts
* Currently enrolled in a clinical trial
* Inability to give informed consent

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward E. Messing, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tamsulosin Group: Subjects will receive:
  1. 0.4mg tamsulosin by mouth nightly for 3 doses prior to the day of surgery and for 2 doses following surgery
  2. education about signs and symptoms of urinary retention
  Tamsulosin: Tamsulosin may have prophylactic properties against post-operative urinary retention
  Education: Education about signs and symptoms of urinary retention
- Education Group: Subjects will receive:
  1) education about signs and symptoms of urinary retention
  Education: Education about signs and symptoms of urinary retention
Period: Overall Study
Arm/Group | Tamsulosin Group | Education Group
Started | 1 | 4
Completed | 1 | 3
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamsulosin Group | Education Group | Total
Number analyzed (Participants) | 1 | 4 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 3
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-operative Urinary Retention
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin Group | Education Group
Number analyzed (Participants) | 1 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Tamsulosin Group | Education Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT02684344/Prot_SAP_000.pdf